CLINICAL TRIAL: NCT02967835
Title: Pilot to Assess Effectiveness of and Satisfaction With Brief Synchronous Tele-psychiatry Consult
Brief Title: Effectiveness and Satisfaction With Brief Synchronous Tele-psychiatry Consult
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: not able to recruit
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mohit Chauhan, M.B.B.S., Senior Associate Consultant, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-003068
Record Dates: First submitted 2016-09-12; First posted 2016-11-18 (Estimated); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Telepsychiatry Consult (Experimental): One time tele-psychiatry consultation to provide treatment recommendations for patients primary care physician.
  Interventions: Behavioral: Tele-psychiatry consult

INTERVENTIONS:
Behavioral: Tele-psychiatry consult — tele-psychiatry consult for evaluation and treatment recommendations

SUMMARY:
Will Tele-psychiatry be effective and acceptable to patients.

DETAILED DESCRIPTION:
This pilot aims to provide tele-psychiatry consults to patients at regional Mayo Clinic Florida primary care sites. The primary aim of this study is to assess the impact of brief tele-psychiatry consults on depression and anxiety outcomes for patients enrolled in complex care management; the secondary aim is to assess patient satisfaction with brief tele-psychiatry consults.

ELIGIBILITY:
Inclusion Criteria

1. Enrolled in complex care management
2. PHQ9 above 10 or GAD7 above 10.

Exclusion Criteria

1. Not able to provide informed consent
2. Severe cognitive impairments or sensory deficits
3. Not able to understand and speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-14 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
Depression Outcome | 6 month
  Will measure depression outcome by measuring PHQ9 score at baseline and 6 months after initial tele-psychiatry consult.
Anxiety Outcome | 6 month
  Will measure Anxiety outcome by using GAD7 score at baseline and 6 months after initial tele-psychiatry consult.

SECONDARY OUTCOMES:
Patient satisfaction with tele-psychiatry consult | baseline visit
  Assess patient satisfaction with tele-psychiatry consult at baseline visit by use of patient satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Chauhan, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No